CLINICAL TRIAL: NCT06560034
Title: VicorderCS NIBP Validation Study to Assess Its Ability to Capture Blood Pressure Measurements
Brief Title: VicorderCS NIBP Validation Study to Review The Ability to Capture Blood Pressure Measurements
Status: Recruiting | Type: Observational
Sponsor: 80 Beats Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00080976
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases; Blood Pressure; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross-Sectional Group: Blood pressure reading of one group of participants
  Interventions: Device: VicorderCS

INTERVENTIONS:
Device: VicorderCS — 1. Vascular Sensor (VCS-VAS-1000) measurement device used with accessories (cuffs and tubes) connected to the device;
  2. Data Station (VCS-DAT-1000) for data collection and analysis

SUMMARY:
80 Beats Medical introduces the VicorderCS, the next generation of our Vicorder technology designed to manage hypertension and cardiovascular risks. This advanced diagnostic equipment offers non-invasive collection and computation of a plethora of cardiovascular markers. It is faster, easier to use, and more portable than its predecessor, with enhanced connectivity options for extended marker collection and analysis. These markers enable early diagnosis of cardiovascular disease, ensuring positive patient outcomes. With a strong foundation in numerous published clinical studies, the VicorderCS enhances data collection and analysis capabilities, empowering the research community in developing new drugs and therapeutics. This validation study is purposed to evaluate one of the physiological parameters that is measured by the VicorderCS system, which is Non-invasive Blood Pressure (NIBP) via the common oscillometric cuff-based method.

DETAILED DESCRIPTION:
The VicorderCS will enable medical personnel to conduct Blood Pressure measurement procedures for the evaluation of a participant's cardiovascular health.

Clinical Rationale This study will compare the accuracy of the 80 Beats Medical noninvasive blood pressure measurement using the VicorderCS device with that of human observers' readings using the auscultatory method, as required by the applicable ISO standard: Non-invasive sphygmomanometers part 2 - clinical investigation of intermittent automated measurement type1. The study will aim to enroll 120 participants for blood pressure readings using both the VicorderCS and auscultatory method using a calibrated aneroid sphygmomanometer.

Design Rationale The VicorderCS blood pressure study will be conducted using consenting participants in Summit County Colorado and designed to be compliant with the requirements within the applicable ISO standard1. Study data, including systolic and diastolic blood pressure readings, will be collected using both the VicorderCS and auscultatory method using a sphygmo-manometer.

Proposed Solution 80 Beats Medical has developed the VicorderCS, which is indicated for the non-invasive measurement of blood pressure to detect cardiovascular health risks.

Device Description

VicorderCS consists of the following components:

1. Vascular Sensor (VCS-VAS-1000) measurement device used with accessories (cuffs and tubes) connected to the device;
2. Data Station (VCS-DAT-1000) for data collection and analysis

Platform Data Privacy and Security The VicorderCS application follows industry best practices for data privacy and security, including compliance with applicable laws and regulations such as the General Data Protection Regulation (GDPR) and the Health Insurance Portability and Accountability Act (HIPAA). 80 Beats Medical has implemented technical and organizational measures to safeguard user data against unauthorized access, disclosure, alteration, or destruction, and regularly conducts security audits and risk assessments to identify and mitigate potential threats.

80 Beats Medical has established policies and procedures to ensure that user data is used only for its intended purpose and is not shared with unauthorized parties.

There are two data sets that will be recorded during this study. One is the pressure waveforms on all four limbs and the other is the Systolic and Diastolic blood pressure measurement on the left arm. All data on the vascular sensor will be deleted after the test is complete. However, the pressure waveforms will be uploaded to the data station before being deleted. This will be part of an internal data pool for use in perpetuity.

Users are provided with transparency and control over their data, including the ability to access, correct, and delete their information. Users can opt out of data collection and sharing, where applicable. Security and privacy of user data are critical to maintaining user trust, and 80 Beats Medical is committed to ensuring the application meets the highest standards for data privacy and security.

STUDY OBJECTIVES Primary Objective The objective of this study is to collect blood pressure readings using the VicorderCS device. We will subsequently conduct statistical analysis by comparing to the traditional sphygmomanometer method according to the ISO standard.

Secondary Objectives A secondary objective of this study is to collect raw waveform data on the opposite arm, and both ankles in order to optimize analysis capabilities in the future.

INVESTIGATIONAL PLAN General Schema of Study Design In this cross-sectional study, we will look at the systolic (Sys) and diastolic (Dia) blood pressure of 120 subjects (ages 18 years or older).

The primary hypothesis of this study is that the VicorderCS can detect and analyze blood pressure in an easy-to-use and portable device providing more complete diagnostics at the point of care.

Study Device 80 Beats Medical has developed the VicorderCSCS, which is indicated for the non-invasive measurement of blood pressure.

Indications for use The VicorderCS Device is indicated for adult patients needing a blood pressure reading.

ELIGIBILITY:
Inclusion Criteria:

* Any gender, in good general health
* Must be 18 years old or older, inclusive at enrollment
* Must be willing to provide blood pressure measurement
* Must be able to read, understand, and willingly sign an Informed Consent Form
* Must be able to read, speak and understand English
* Must be available to attend one study visit at: please specify exact location.

Exclusion Criteria:

* Excluding subjects with significantly irregular heart rhythm (e.g. Bigeminy, trigeminy, isolated ventricular premature beat (VPB), atrial fibrillation) or are pregnant
* No active email address
* Non-English or Spanish- speaking
* Unable to read in English.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy individuals meeting inclusion criteria in the Colorado area
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Reading | One visit (1hour)
  Collect blood pressure readings using the VicorderCS device

SECONDARY OUTCOMES:
Waveform Data | One visit (1hour)
  Collect raw waveform data on the opposite arm, and both ankles in order to optimize analysis capabilities in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Vaswani, MD, Principal Investigator — PI
Locations (1):
- Manos Health Study Site, Breckenridge, Colorado, United States

IPD SHARING:
Plan to Share IPD: No